CLINICAL TRIAL: NCT07404098
Title: Efficacy Of Eggshell-Derived Nanohydroxyapatite Based Mineralized Plasmatic Matrix Versus Xenogeneic Based Mineralized Plasmatic Matrix in Posterior Mandibular Socket Preservation: A Randomized Controlled Clinical Trial.
Brief Title: Efficacy Of Eggshell-Derived Nanohydroxyapatite Based Mineralized Plasmatic Matrix Versus Xenogeneic Based Mineralized Plasmatic Matrix in Posterior Mandibular Socket Preservation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammad Fardous Alfardous Alazm, Principal Investigator Mohammad Fardous, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: per3322026
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: Alveolar Bone Resorption; Socket Preservation; Wound Healing; Nano-hydroxyapatite
Keywords: bone gain; xenograft; EnHa; socket preservation; prf
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eggshell-derived nanohydroxyapatite-based mineralized plasmatic matrix along with PRF (Experimental): A whole venous blood (10 ml) is obtained from the patient to prepare the PRF. The 10 ml are divided into: 5 ml for mixing and 5 ml to be used as a covering membrane.
  Tooth extraction is done comprising minimal surgical trauma to the surrounding bone using periotomes and remaining root forceps. Then, debriding the socket using bone curette will be done.
  PRF will be prepared as instructed by (Choukroun et al., 2006) the first (5 ml) of PRF will be mixed with the eggshell nanohydroxyapatite- based matrix (EnHA) and it will be placed inside the socket.
  The second (5ml) of PRF will be used as a membrane. The suturable membrane formation is prepared from fibrin clot by pressing it in PRF Box.
  Primary closure is done by appropriate suturing technique (Criss Cross Suture/ Figure of 8.) by using resorbable suture material (Vicryl).
  Interventions: Procedure: Socket preservation using eggshell-derived nanohydroxyapatite-based mineralized plasmatic matrix along with platelet-rich fibrin (PRF).
- deproteinized bovine bone mineral (DBBM) xenograft along with platelet-rich fibrin (PRF). (Active Comparator): A whole venous blood (10 ml) is obtained from the patient to prepare the PRF. The 10 ml are divided into: 5 ml for mixing and 5 ml to be used as a covering membrane.
  Tooth extraction is done comprising minimal surgical trauma to the surrounding bone using periotomes and remaining root forceps. Then, debriding the socket using bone curette will be done.
  PRF will be prepared as instructed by (Choukroun et al., 2006) the first (5 ml) of PRF will be mixed with Deproteinized Bovine Bone Mineral (DBBM) and it will be placed inside the socket.
  The second (5ml) of PRF will be used as a membrane. The suturable membrane formation is prepared from fibrin clot by pressing it in PRF Box.
  Primary closure is done by appropriate suturing technique (Criss Cross Suture/ Figure of 8.) by using resorbable suture material (Vicryl).
  Interventions: Procedure: Socket preservation using deproteinized bovine bone mineral (DBBM) xenograft along with platelet-rich fibrin (PRF).

INTERVENTIONS:
Procedure: Socket preservation using eggshell-derived nanohydroxyapatite-based mineralized plasmatic matrix along with platelet-rich fibrin (PRF). — A whole venous blood (10 ml) is obtained from the patient to prepare the PRF. The 10 ml are divided into: 5 ml for mixing and 5 ml to be used as a covering membrane.
  Tooth extraction is done comprising minimal surgical trauma to the surrounding bone using periotomes and remaining root forceps. Then, debriding the socket using bone curette will be done.
  PRF will be prepared as instructed by (Choukroun et al., 2006) The Blood is obtained from the patient and centrifuged for 3000rpm for 10 min The first (5 ml) of PRF will be mixed with the eggshell nanohydroxyapatite- based matrix (EnHA) and it will be placed inside the socket.
  The second (5ml) of PRF will be used as a membrane. The suturable membrane formation is prepared from fibrin clot by pressing it in PRF Box.
  Primary closure is done by appropriate suturing technique (Criss Cross Suture/ Figure of 8.)by using resorbable suture material (Vicryl).
  Arms: eggshell-derived nanohydroxyapatite-based mineralized plasmatic matrix along with PRF
Procedure: Socket preservation using deproteinized bovine bone mineral (DBBM) xenograft along with platelet-rich fibrin (PRF). — A whole venous blood (10 ml) is obtained from the patient to prepare the PRF. The 10 ml are divided into: 5 ml for mixing and 5 ml to be used as a covering membrane.
  Tooth extraction is done comprising minimal surgical trauma to the surrounding bone using periotomes and remaining root forceps. Then, debriding the socket using bone curette will be done.
  PRF will be prepared as instructed by (Choukroun et al., 2006) The Blood is obtained from the patient and centrifuged for 3000rpm for 10 min. The first (5 ml) of PRF will be mixed with Deproteinized Bovine Bone Mineral (DBBM) and it will be placed inside the socket.
  The second (5ml) of PRF will be used as a membrane. The suturable membrane formation is prepared from fibrin clot by pressing it in PRF Box.
  Primary closure is done by appropriate suturing technique (Criss Cross Suture/ Figure of 8.) by using resorbable suture material (Vicryl).
  Arms: deproteinized bovine bone mineral (DBBM) xenograft along with platelet-rich fibrin (PRF).

SUMMARY:
After tooth extraction, the alveolar bone, which supports the teeth, undergoes a natural resorption process. This bone loss can be significant, especially in the first few months post-extraction, leading to a reduction in both bone height and width (Araújo et al ,. 2005) Generally, the goal of alveolar ridge preservation is to maximize bone formation while maintaining good soft tissue architecture, As socket preservation has proved high clinical efficacy in maintaining alveolar ridge high and width, there are many materials that have been proposed such as: autogenous bone grafts, allografts, xenografts, alloplasts, dentin graft and PRF. Unfortunately, the previously mentioned grafting material has several limitations have more such as high cost, biocompatibility, osteoinductive limitations and the need for a second surgical site. These limitations encouraged the researchers to test alternative materials and techniques to provide comparable or superior outcomes with fewer drawbacks.

One of the newly introduced materials is eggshell derived nanohydroxyapatite (EnHA). Eggshell-derived nanohydroxyapatite (EnHa) represents a novel and potentially superior alternative due to its biocompatible, osteoconductive, and osteoinductive bone substitute. Preliminary studies suggest that this material.

The synergistic effect of PRF when combined with various graft materials has also been extensively studied. when PR combined with bone grafting materials, it results in enhanced osteoconductive properties of graft materials and promotes efficient bone regeneration. (Yilmaz et al., 2017).

However, up till now, there are no sufficient studies on the clinical efficacy of EnHA as a cheaper and readily available alternative which has superior clinical properties especially when combined with PRF compared to standard xenografts.

DETAILED DESCRIPTION:
After tooth extraction, the alveolar bone, which supports the teeth, undergoes a natural resorption process. This bone loss can be significant, especially in the first few months post-extraction, leading to a reduction in both bone height and width (Araújo et al., 2005). This resorption can compromise the structural foundation required for future dental restorations, such as implants, bridges, or dentures.

Maintaining the alveolar ridge's volume and contour is crucial for the successful placement of dental implants. Adequate bone volume ensures that implants can be securely anchored, providing the necessary stability and support for prosthetic teeth (Jung et al., 2013). Without sufficient bone, additional procedures such as bone grafting may be required, which can increase treatment time, cost, and patient discomfort. Bone loss can lead to changes in the facial structure, such as sunken cheeks and lips, which can affect a patient's appearance and self-esteem.

By preserving the socket, dental professionals can help maintain the natural contour of the jawline and facial aesthetics (Schropp et al., 2003).

Socket preservation can reduce the risk of complications associated with bone loss, such as the migration of adjacent teeth, changes in occlusion, and the development of periodontal pockets. These complications can lead to further dental issues and complicate future restorative procedures (Ten Heggeler et al., 2011).

The use of appropriate materials in socket preservation can promote bone regeneration and soft tissue healing, leading to better clinical outcomes and patient satisfaction (Vignoletti et al., 2012).

Traditional methods for socket preservation have been developed to address the challenges associated with alveolar ridge resorption following tooth extraction. These methods primarily focus on using various grafting materials and techniques to maintain the socket's volume and promote bone regeneration.

Autogenous bone grafts involve harvesting bone from the patient's own body, typically from intraoral sites such as the mandibular ramus or chin. These grafts are considered the gold standard due to their osteogenic, osteoinductive, and osteoconductive properties. However, the need for a secondary surgical site increases patient morbidity and the complexity of the procedure. (Schwarz et al., 2012).

Allografts sourced from human donors and processed for sterilization, such a demineralized freeze-dried bone allograft (DFDBA), had been used for their osteoinductive properties and availability, significantly reducing ridge resorption compared to normal healing procedure and socket preservation (Iasella et al., 2003).

xenogeneic graft materials such as deproteinized bovine bone mineral (DBBM), are widely used in socket preservation. These materials are derived from animal sources and undergo extensive processing to remove organic components leaving behind a mineral matrix that is highly osteoconductive. DBBM, for example, has been shown to support new bone formation and maintain ridge dimensions effectively (Araújo et al., 2009). Despite their effectiveness, xenogeneic materials can be expensive and may raise concerns about biocompatibility and disease transmission.

Alloplastic materials are synthetic bone substitutes, such as hydroxyapatite, tricalcium phosphate, and bioactive glass. These materials are designed to mimic the mineral component of natural bone and provide a scaffold for new bone growth. Alloplastic materials are biocompatible and eliminate the risk of disease transmission. However, their properties may be limited compared to natural bone grafts (Jung et al., 2013).

Eggshell-derived nanohydroxyapatite (EnHA) represents a novel and promising material for guided bone regeneration and socket preservation. This material is derived from natural eggshells, which are primarily composed of calcium carbonate (CaCO3). Through a series of chemical processes, the calcium carbonate in eggshells can be converted into nanohydroxyapatite, a form of calcium phosphate that closely resembles the mineral component of human bone. Here are the key aspects and benefits of using eggshell-derived nanohydroxyapatite in socket preservation: First, its excellent biocompatibility. This biocompatibility ensures that the material integrates well with the surrounding natural bone tissue, promoting bone healing and regeneration. (Ramesh et al., 2018).

Eggshell-derived nanohydroxyapatite provides a scaffold that supports the attachment, proliferation, and differentiation of osteoblasts, the cells responsible for bone formation. This osteoconductive property is crucial for effective bone regeneration, as it facilitates the growth of new bone tissue within the socket (Sivolella et al., 2012).

Eggshells are an abundant and inexpensive byproduct of food industry, making them a more readily available and cost-effective alternative for ridge preservation. This cost-effectiveness makes socket preservation procedures utilizing (EnHA) a cheaper and effective option for many patients. (Ramesh et al., 2018).

Utilizing eggshells to produce nanohydroxyapatite also addresses environmental concerns. By recycling waste materials from the food industry, this approach contributes to waste reduction and promotes sustainable practices in biomaterial production (Ramesh et al., 2018).

Nanohydroxyapatite derived from eggshells exhibits enhanced mechanical properties compared to other forms of hydroxyapatite. The nanoscale particles provide a larger surface area, which can improve the material's strength and durability. These properties are essential for maintaining the structural integrity of the socket during the healing process (Sivolella et al., 2012).

Many studies have demonstrated the potential of eggshell-derived nanohydroxyapatite in promoting bone regeneration and socket preservation. In 2012, Sivolella et al. reported EnHA new bone formation with histological evidence of osteointegration. However, they recommended more extensive clinical trials to validate these findings and establish standardized protocols for its use in dental practice. Clinical and radiographic assessments are essential for evaluating the efficacy of socket preservation materials. These assessments provide insights into bone density, volume maintenance, and overall healing outcomes. Studies have shown that both clinical and radiographic evaluations are crucial for determining the success of socket preservation techniques (Jung et al., 2013).

Several studies have demonstrated the efficacy of PRF in socket preservation following tooth extraction. A randomized controlled trial by Temmerman et al. (2016) evaluated the use of PRF

in preserving alveolar ridge dimensions post-extraction. This study found that PRF significantly reduced the vertical and horizontal bone loss compared to the control group, which did not receive PRF. The authors concluded that PRF could effectively enhance soft tissue healing and maintain ridge dimensions, making it a valuable tool in socket preservation.

Moreover, the synergistic effect of PRF when combined with various graft materials has also been extensively studied. A study by Choukroun et al. (2006) investigated the combination of PRF with deproteinized bovine bone mineral (DBBM) for sinus lift procedures. The results showed that the combination of PRF and DBBM led to enhanced bone formation and faster healing compared to DBBM alone. This finding suggests that PRF can enhance the osteoconductive properties of graft materials, promoting more efficient bone regeneration.

Clinical and radiographic outcomes are critical in assessing the efficacy of PRF in socket preservation. A systematic review by Miron et al. (2017) analyzed various studies on PRF and concluded that PRF consistently improved soft tissue healing, reduced postoperative pain and swelling, and enhance bone regeneration. Additionally, radiographic evaluations showed increased bone density and volume in sites treated with PRF.

Despite these promising results, of the up mentioned studies the preliminary findings showed a gap of knowledge regarding the efficacy of eggshell-derived nanohydroxyapatite-based matrices along with platelet-rich fibrin (PRF) to traditional xenogeneic-based matrices. These further studies are necessary to provide robust evidence and guide clinical decision-making (Jensen et al., 2014).

This research aims to address this gap by conducting a randomized controlled clinical trial to evaluate and compare the clinical and radiographic outcomes of these two materials in posterior mandibular socket preservation.

Choice of Comparators:

Based on what had been mentioned previously randomized controlled clinical trial, the efficacy of eggshell-derived nanohydroxyapatite-based (EnHA) along with platelet-rich fibrin (PRF) will be compared to deproteinized bovine bone mineral (DBBM) along with platelet-rich fibrin (PRF) for posterior mandibular socket preservation. DBBM is chosen as the comparator due to its availability use and well-documented success in maintaining alveolar ridge dimensions and supporting new bone formation (Araújo & Lindhe, 2009). Known for its osteoconductive properties, DBBM serves as a standard reference material, providing a robust benchmark for evaluating the performance of the eggshell-derived nanohydroxyapatite-based matrix. This comparison aims to determine if the novel eggshell-derived matrix offers comparable or superior outcomes in terms of bone regeneration, ridge preservation, and overall clinical success, thereby potentially offering a more cost-effective and sustainable alternative for socket preservation.

The preservation of alveolar ridge dimensions following tooth extraction is essential for the success of subsequent dental restorations. Traditional graft materials, such as xenogeneic-based mineralized matrices, have been widely used either alone or in combination with Platelet-Rich Fibrin (PRF) to enhance bone regeneration and soft tissue healing. However, these materials may have limitations, including potential immunogenic responses and variable integration (Temmerman et al., 2016).

Eggshell-derived nanohydroxyapatite (EnHa) represents a novel and potentially superior alternative due to its biocompatible, osteoconductive, and osteoinductive bone substitute. Preliminary studies suggest that this material, when combined with PRF, may enhance bone regeneration and maintain alveolar ridge dimensions more effectively than traditional xenogeneic-based matrices (Yilmaz et al., 2017).

This research is being proposed to fill the gap on knowledge clinical and radiographic data on the clinical efficacy of these two grafting approaches. By evaluating the outcomes in a randomized controlled clinical trial, this study aims to determine clinically and radiographically whether the eggshell-derived nanohydroxyapatite-based matrix with PRF offers superior benefits in terms of bone quality, volume preservation, and overall clinical success with low financial efforts. (Miron et al., 2017).

ELIGIBILITY:
* Inclusion criteria:

  1. Patient having at least one hopeless posterior mandibular tooth requires extracted
  2. 18 years old or older.
  3. Non- smoker
  4. Motivated patients with good enough understanding of oral health measurements and importance
  5. Medically fit patients.
  6. No acute infections, pus formation, socket and bony discharges.
  7. Compliant the patient to ensure the follow up
* Exclusion criteria:

  1. Heavy smokers (more than 10 cigarettes per day or an electronic cigarette dose of >6 mg/ml of nicotine).
  2. Pregnant subjects.
  3. Presence of active infection or severe inflammation in the intervention zone.
  4. Relevant medical history contraindicates implant surgery.
  5. Immunosuppression (e.g.: HIV, solid-organ transplants).
  6. Head and neck-irradiated patients in the past 5 years.
  7. Regular intake of bisphosphonates, anticoagulants as: aspirin, or anti-inflammatories.
  8. Patients with anemia or Thrombocytopenia.
  9. Chronic drug abuse or alcoholic habits.
  10. Patients with poor oral hygiene (full-mouth plaque score and full-mouth bleeding score >15%) and lack of motivation.
  11. Uncontrolled diabetes (reported levels of glycated hemoglobin exceeding 7%).
  12. Uncontrolled and /or untreated periodontal disease (Active Periodontitis).
  13. Patients with significant comorbidity such as recent heart attack or coagulation disorder.
  14. Patients with a history of allergies.
  15. Mentally and physically handicapped patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in bone density | after 4 months postoperatively.
  CBCT scans will be performed at baseline and 4 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. Bone density measured using CBCT radiographs after 4 months later, and a 12*12 mm² region of measurement used to assess the density in different points (Point A at the socket crest, Point B at the middle of the socket, Point C at the apex). The CBCT taken after 4 months will serve the purpose of superimposing the two scans and assessing the bone density changes after augmentation. These measurements will be denoted as HW-1, HW-3, and HW-5, respectively.

SECONDARY OUTCOMES:
Percentage of new vital bone formation | After 4 months postoperatively
  The biopsies will be stored in a 10% formalin solution for preservation. Afterward, they will undergo decalcification in EDTA for a duration of four weeks. Following decalcification, the specimens will be processed and embedded in paraffin to create tissue blocks. Longitudinal sections of 5μm thickness will be cut from the paraffin blocks. These sections will be stained using hematoxylin and eosin (H&E) or Masson's trichromatic (MT) stains for histological evaluation and histomorphometry analysis. Photomicrographs of the stained sections will be captured using a digital light microscope (Leica Digital Microscope, Leica Microsystems, Germany).
  Histomorphometry analysis will be performed to quantify the area percentage occupied by bone, graft particles, and soft tissue stroma relative to the total examined histological area. Image analyzer software (Leica QWin 500 image analysis software, Leica Microsystems, Switzerland) will be used for this analysis.
Change in Percentage of residual bone graft | after 4 months postoperatively
  CBCT scans will be performed at baseline and 4 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish a reference, the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn. The vertical reference line will be placed at the midpoint of the extraction socket, intersecting the apical reference point.
  The height of the alveolus will be measured at the mid-buccal aspect (BH) and mid-lingual aspect (LH).
Wound healing and pain | 10 days post operative and after 4 months postoperative
  Scale out of 7 points according to Modified healing index (MHI) (Pippi et al..2013)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Darhous, Professor, Study Director — Cairo University; Mohammed Fardous Alfardous AlAzm, Bachelor, Principal Investigator — Cairo University; Maie Esmaiel, Lecturer, Study Chair — Cairo University; Mohamed Omara, Associate Professor, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt